CLINICAL TRIAL: NCT05901870
Title: Russian National Health Telephone Survey (RNHTS): Health-Related Quality of Life, Health-Related Behaviors, Health Care Utilization
Brief Title: Russian National Health Telephone Survey (RNHTS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Agency of Social Information St. Petersburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: 03.005.С.34.1
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-06

CONDITIONS: Public Health
Keywords: health status; health-related quality of life; health-related behaviors; health care utilization; telephone survey; national health survey
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Russian Adults (18+): Russian adults who meet the inclusion criteria (described below) will be participants of RNHTS.
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — All study participants will be surveyed with the questionnaire, which includes such instruments as EQ-5D-3L and WG-SS, to assess their health-related quality of life, health-related behavior, and health care utilization indicators.

SUMMARY:
Russian National Health Telephone Survey (RNHTS) is a public health surveillance study that assesses various health-related quality of life, health-related behavior, and health care utilization indicators on a representative sample of the adult Russian population. All data will be collected via a Computer Assisted Telephone Interview (CATI).

DETAILED DESCRIPTION:
Russian National Health Telephone Survey (RNHTS) is the first public health surveillance study in Russia. The aim of RNTHS is to obtain unique representative data on health-related quality of life, health-related behaviors, and health care utilization indicators for the adult Russian population. Analysis of these indicators provides a detailed outlook on how health is associated with people's well-being, quality of life, and socio-demographic characteristics, which adds to official and aggregated statistics for Russia.

RNHTS consists of five sections. Section 1 includes socio-demographic characteristics of respondents such as their gender, age, marital status, education level, income level, employment status and location. Section 2 measures indicators of general health and health-related quality of life using the 3-level version of the EuroQol-5 Dimension questionnaire (EQ-5D-3L) and the Washington Group Short Set on Functioning questionnaire (WG-SS). Section 3 covers three health-related behaviours of respondents: smoking, drinking alcohol, and physical activity. Section 4 consists of questions about health care utilization in the last 12 months with an emphasis on patient choice between public and private health care. This section also measures how satisfied respondents were with health care services that they used, their unmet needs, and their health care avoidance. Section 5 is modifiable for each round (year) of RNHTS. This version of the protocol describes round 2 of RNHTS. In this round, Section 5 is devoted to measuring prevalence of arthritis in the adult Russian population and how it affects their quality of life as well as to learning about oral health and dental services utilization among Russian adults.

More than 2000 respondents will be randomly selected for RNHTS. All data will be collected using a Computer Assisted Telephone Interview (CATI) system, which allows real-time data capture and consolidation. All interviews will be conducted anonymously. The telephone survey will be conducted by Agency of Social Information St. Petersburg (ASI St. Petersburg). RNHTS data will be analysed using statistical analysis methods which will be presented using summary tables (summary statistics, contingency tables, frequency distributions), correlation coefficients, and estimates of regression models (coefficients, odds ratios, marginal effects). The results of statistical analysis will be compiled in one report with authors' comments on the findings.

ELIGIBILITY:
Inclusion Criteria:

* Respondents are aged 18 and above.
* Respondents provide informed consent via telephone at the beginning of the survey.

Exclusion Criteria:

* Respondents refuse to provide informed consent.
* Respondents are severely ill or too frail to participate.
* Respondents have cognitive problems.
* Respondents have hearing or speaking problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult Russian residents are eligible for the survey.
Sampling Method: Probability Sample
Enrollment: 2529 (Actual)
Dates: Start 2023-08-12 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Self-assessed health status | Upon enrollment
  Respondents will be asked to rate their health with the "in general, would you say that your health is excellent, very good, good, fair, or poor?" question. The answer that they choose represents their self-assessed (self-rated) health status.
Quality of life indicator measured by the 3-level version of the EuroQol-5 Dimension questionnaire (EQ-5D-3L) - health profile (state) | Upon enrollment
  The EQ-5D-3L questionnaire consists of 5 questions in 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In the 3-level version of the questionnaire, each domain has 3 levels. The 5 answers to the 5 questions are combined into a 5-digit number that describes the patients' health profile (state).
The visual analogue scale score (EQ-VAS) | Upon enrollment
  The EQ-VAS records the patients' self rated-health on a scale from 0 to 100, where 0 = the worst imaginable health and 100 = the best imaginable health.
Disability and functional limitations according to the Washington Group Short Set on Functioning questionnaire (WG-SS) | Upon enrollment
  The WG-SS questionnaire is comprised of 6 questions about 6 core functional domains: seeing, hearing, walking, cognition, self-care, and communication. Each question has four response categories: " no difficulty", " some difficulty", "a lot of difficulty", "cannot do it at all". Disability is identified for individuals whose answer to at least one of the questions is "have a lot of difficulty" or "cannot do at all". Presence of functional limitations is also determined within each domain for each person if their answer to a question about the domain is either "have a lot of difficulty" or "cannot do at all".
Body Mass Index (BMI) | Upon enrollment
  Self-reported height (in meters) and self-reported weight (in kilograms) will be combined to measure BMI as a person's weight divided by the square of their height.
Smoking behaviour | Upon enrollment
  Respondents will be asked whether they are current smokers or not, and if so, they will be questioned about smoking devices they use, their smoking frequency, intensity of smoking, smoking history and intentions to quit smoking.
Alcohol consumption | Upon enrollment
  Respondents will be asked whether they consume alcoholic beverages or not, and if so, they will be asked about the volume of consumed alcoholic beverages.
Physical activity | Upon enrollment
  The frequency of physical activity and sedentary time will cover the physical activity section.
Health care utilisation and patient choice between public and private health care providers | Upon enrollment
  Respondents will be asked whether they visited a health care provider in the last 12 months. They will be asked to specify whether they chose to go to a public health care provider, to a private health care provider or whether they went to both types of providers.
Satisfaction with health care services provided | Upon enrollment
  Respondents will be asked 4 questions about their satisfaction with their most recent visit to a health care provider in the last 12 months. They will be asked to rate how clear their doctor's explanation of their health problem was on a 5-level scale, how clear the doctor's explanation of their treatment options was on a 5-level scale, whether they trusted their doctor (fully trusted, partially trusted, or did not trust at all), and whether they would choose to get the same health care service at the same facility again if they had to (yes/no question).
Nonreceipt of needed medical care and nonreceipt of needed prescription drugs | Upon enrollment
  This outcome measure refers to three types of cases of unmet needs:
  * Respondents will be surveyed about cases when they went to a health care provider but were refused services. If respondents report that such an instance occurred in the last 12 months, they will be asked to specify the reason for the refusal that they were given.
  * Respondents will also be asked whether they wanted to seek help for some health problem but ultimately decided not to in the last 12 months. If respondents report deciding not to seek care, they will be asked to specify the reasons that guided their decision.
  * Respondents will also be asked whether they were prescribed some medication but ultimately decided not to buy it in the last 12 months. If respondents report deciding not to buy prescribed drugs, they will be asked to specify the reasons that guided their decision.

SECONDARY OUTCOMES:
Oral health | Upon enrollment
  Respondents will be asked to rate their oral health with the "in general, would you say that your oral health is excellent, very good, good, fair, or poor?" question. Respondents will also be questioned about practices they use for healthy teeth and gums.
Dental services utilisation | Upon enrollment
  Respondents will be asked when they last visited a dental care practitioner. They will be asked to specify where they chose to go: to a public dental care practitioner or to a private dental care practitioner. Respondents will be asked whether they wanted to seek help for dental problems but ultimately decided not to go to a dental care practitioner in the last 12 months. If respondents report deciding not to seek dental care, they will be asked to specify the reasons that guided their decision.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Aleksandrova, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No